CLINICAL TRIAL: NCT00808470
Title: Micronutrient Intervention to Reduce Noise-Induced Hearing Loss: Prevention of Temporary Threshold Changes Induced by Use of a Digital Music Player
Brief Title: Micronutrients to Prevent Noise-induced Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Florida (Other); Southern Illinois University (Other); Hearing Health Science, Inc. (Unknown)
Responsible Party: Principal Investigator, Glenn Green, Associate Professor of Otolaryngology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01DC008423 (NIH); U01DC008423-02S1 (NIH); U01DC008423-03 (NIH); U01DC008423 (NIH)
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Noise-Induced Hearing Loss
Keywords: Noise; Hearing Loss; Tinnitus; Antioxidant; Vasodilator; Beta-Carotene; Vitamin C; Vitamin E; Magnesium
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Hearing Loss; Tinnitus | interventions — beta Carotene; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrients (Experimental): Subjects in University of Florida music player study who are assigned to nutrient condition(beta-carotene, vitamins C and E, magnesium). Nutrient tablets are consumed for 4 days.
  Interventions: Drug: beta-carotene, vitamins C and E, magnesium
- Placebo for nutrients (Placebo Comparator): Subjects in University of Florida music player study who are assigned to control (placebo) condition. Placebo tablets are consumed for 4 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: beta-carotene, vitamins C and E, magnesium — 6 mint-flavored tablets per day, taken once daily
  total daily dose label claim: micronutrient combination of 500 mg vitamin C (magnesium ascorbate), 315 mg magnesium (magnesium citrate, magnesium ascorbate, magnesium stearate), 267 mg vitamin E (d-α-tocopherol acetate), and 18 mg beta carotene.
  Other Names: Soundbites®
  Arms: Nutrients
Other: Placebo — 6 mint-flavored tablets per day, containing inactive substances including mannitol, peppermint flavor, sucralose, color prep, iron oxide yellow synthetic, stearic acid (vegetable grade), and silicon dioxide colloidal.
  Arms: Placebo for nutrients

SUMMARY:
Noise-induced hearing loss (NIHL) is a significant clinical, social, and economic issue. Studies in animals have allowed us to identify mechanisms contributing to NIHL, including direct mechanical trauma, free radicals formed in association with metabolic stress, and reduced blood flow. A combination of antioxidant vitamins (beta-carotene, and vitamins C and E) and the mineral magnesium (which acts in part as a vasodilator but also as an antioxidant) is highly effective in preventing NIHL in animals. These studies evaluate efficacy of this intervention in humans.

Hypothesis: Treatment with these micronutrients provides safe, effective attenuation of acute hearing changes induced by exposure to real-world sounds producing temporary (non-permanent) or permanent hearing changes induced by exposure to real-world sounds.

Experiment 1: "Digital Audio Player" studies (University of Florida, Gainesville). Prevention of *temporary* elevations in hearing thresholds, induced by exposure to moderately loud music, will be measured. Subjects will be 70 young adults with equal numbers of male and female participants.

DETAILED DESCRIPTION:
This study assessed the potential for prevention of the temporary changes in hearing that can occur after use of a music player device for 4 hours. All participants listened to one of two playlists (pop or rock) set at the same volumes to provide equivalent and consistent exposures across participants. Participants received either a dietary supplement or a placebo once/daily for three days prior to the day of music exposure, and also on the day of music exposure. The fourth and final dose was consumed immediately prior to music listening and consumption was observed by a member of the study team. Changes in hearing were assessed 15-min post-music, and then 1, 2, and 3 hours later, as well as the following day and 1 week later.

ELIGIBILITY:
Inclusion Criteria:

Hearing inclusion criteria are as follows for all studies:

* subjects must have a normal audiologic assessment at baseline consisting of:

  1. symmetric hearing with air conduction thresholds no worse than 25 dB HL at tested frequencies between .25 - 8 kHz;
  2. no significant threshold asymmetry (i.e., greater than 15 dB) between the ears at any test frequency;
  3. no significant air-bone gaps (i.e., greater than 10 dB); and
  4. Type A tympanograms bilaterally, defined as a range of -140 to +40 daPa based on the 90% range for adults (Margolis & Hunter 2000).

Additional criteria are as follows:

* No history of ear disease, able to provide informed consent, agree to follow study procedures, normal health screening at study entry

Exclusion Criteria:

* Pregnant or trying to become pregnant within study period (females)
* subjects belonging to vulnerable populations
* subjects with any history of chronic disease
* hearing loss that exceeds limits specified above
* inability or failure to provide informed consent
* medical conditions that require treatment with drugs including anticoagulants
* diuretics
* digoxin
* aspirin/salicylate
* barbiturates
* minocycline

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef M Miller, PhD, Principal Investigator — University of Michigan; Colleen G Le Prell, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Le Prell CG, Fulbright A, Spankovich C, Griffiths SK, Lobarinas E, Campbell KC, Antonelli PJ, Green GE, Guire K, Miller JM. Dietary supplement comprised of beta-carotene, vitamin C, vitamin E, and magnesium: failure to prevent music-induced temporary threshold shift. Audiol Neurotol Extra. 2016 May-Aug;6(2):20-39. doi: 10.1159/000446600. Epub 2016 Jul 5. PMID 27990155
- [Result] Le Prell CG, Johnson AC, Lindblad AC, Skjonsberg A, Ulfendahl M, Guire K, Green GE, Campbell KC, Miller JM. Increased vitamin plasma levels in Swedish military personnel treated with nutrients prior to automatic weapon training. Noise Health. 2011 Nov-Dec;13(55):432-43. doi: 10.4103/1463-1741.90317. PMID 22122960
- [Derived] Spankovich C, Le Prell CG. Associations between dietary quality, noise, and hearing: data from the National Health and Nutrition Examination Survey, 1999-2002. Int J Audiol. 2014 Nov;53(11):796-809. doi: 10.3109/14992027.2014.921340. Epub 2014 Jun 30. PMID 24975234
- [Derived] Le Prell CG, Yang Q, Harris JG. Modification of digital music files for use in human temporary threshold shift studies. J Acoust Soc Am. 2011 Oct;130(4):EL142-6. doi: 10.1121/1.3630017. PMID 21974483

RESULTS

PARTICIPANT FLOW:
Groups:
- Nutrients: Dietary Supplement. Subjects in University of Florida music player study who are assigned to active agent treatment group. Nutrient tablet treatments are consumed for 4 days.
  Dietary supplement consisting of beta-carotene, vitamins C and E, magnesium: 6 mint-flavored tablets per day, taken once daily
  total daily dose label claim: micronutrient combination of 500 mg vitamin C (magnesium ascorbate), 315 mg magnesium (magnesium citrate, magnesium ascorbate, magnesium stearate), 267 mg vitamin E (d-α-tocopherol acetate), and 18 mg beta carotene.
- Placebo for Nutrients: Subjects in University of Florida music player study who are assigned to control (placebo) condition. Placebo tablets are consumed for 4 days.
  Placebo Control: 6 mint-flavored tablets per day, containing inactive substances including mannitol, peppermint flavor, sucralose, color prep, iron oxide yellow synthetic, stearic acid (vegetable grade), and silicon dioxide colloidal.
Period: Overall Study
Arm/Group | Nutrients | Placebo for Nutrients
Started | 37 | 35
Completed | 35 | 35
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: healthy young adults that meet audiometric enrollment criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutrients | Placebo for Nutrients | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (2.4) | 21.3 (2.4) | 21.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 25 | 26 | 51
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Average Threshold Shift at 4 kHz in Both Ears
Description: The study measures the quietest decibel level the participants can hear before the 4 hour music exposure The first post-music test to measure shift is 15 minutes after the music exposure is completed and again at 1 hour intervals. The shift represents the mean change in quietest decibel volume detected between baseline (pre-music) and post music.
Time Frame: 15 min, 1 hr intervals for 3 hours to measure temporary changes; additional tests at 1 day and 1 week post-exposure.
Population: All subjects that completed music exposure were analyzed; two subjects withdrew from study prior to music exposure.
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Nutrients | Placebo for Nutrients
Number analyzed (Participants) | 35 | 35
decibels
  15 minutes post exposure | 3.94 (4.39) | 3.4 (3.81)
  1 hour and 15 minutes after exposure | 2.77 (4.00) | 2.03 (3.12)
  2 hours and 15 minutes after exposure | 2.27 (3.81) | 2.03 (3.12)
  3 hours and 15 minutes after exposure | 1.51 (3.18) | .88 (2.48)
  1 day after exposure | .09 (1.91) | .00 (1.91)
  1 week after exposure | -.57 (2.25) | .11 (2.25)
Statistical Analysis 1: Comparison: Nutrients vs Placebo for Nutrients; 15 minutes after exposure; Test type: Superiority or Other; p = 0.58, t-test, 2 sided
Statistical Analysis 2: Comparison: Nutrients vs Placebo for Nutrients; 1 hour and 15 minutes after exposure; Test type: Superiority or Other; p = 0.39, t-test, 2 sided
Statistical Analysis 3: Comparison: Nutrients vs Placebo for Nutrients; 2 Hours 15 minutes after exposure; Test type: Superiority or Other; p = .51, t-test, 2 sided
Statistical Analysis 4: Comparison: Nutrients vs Placebo for Nutrients; 3 hours, 15 minutes after exposure; Test type: Superiority or Other; p = .36, t-test, 2 sided
Statistical Analysis 5: Comparison: Nutrients vs Placebo for Nutrients; 1 day after exposure; Test type: Superiority or Other; p = .86, t-test, 2 sided
Statistical Analysis 6: Comparison: Nutrients; 1 week after exposure; Test type: Superiority or Other; p = .24, t-test, 2 sided

2. Secondary Outcome: Threshold Shift at Individual Frequencies, Including 0.25, 0.5, 1, 2, 3, 6, and 8 kHz, 15 Min Post-music
Description: as for outcome 1
Time Frame: 15 min
Population: all participants that completed music exposure were assessed; two participants withdrew prior to music exposure.
Measure: Mean (Standard Deviation); unit: decibels
Groups:
- Nutrients: Dietary Supplement. Subjects in UF music player study who are assigned to active agent treatment group. Nutrient tablet treatments are consumed for 4 days.
  Dietary supplement consisting of beta-carotene, vitamins C and E, magnesium: 6 mint-flavored tablets per day, taken once daily
  total daily dose label claim: micronutrient combination of 500 mg vitamin C (magnesium ascorbate), 315 mg magnesium (magnesium citrate, magnesium ascorbate, magnesium stearate), 267 mg vitamin E (d-α-tocopherol acetate), and 18 mg beta carotene.
- Placebo for Nutrients: Subjects in UF music player study who are assigned to control (placebo) condition. Placebo tablets are consumed for 4 days.
  Placebo Control: 6 mint-flavored tablets per day, containing inactive substances including mannitol, peppermint flavor, sucralose, color prep, iron oxide yellow synthetic, stearic acid (vegetable grade), and silicon dioxide colloidal.
Arm/Group | Nutrients | Placebo for Nutrients
Number analyzed (Participants) | 35 | 35
decibels
  250 Hz | 0.2571 (0.3487) | 1.2286 (0.4921)
  500 Hz | 0.8 (0.4177) | 1.0000 (0.3932)
  1000 Hz | 1.6571 (0.4119) | 1.6857 (0.4505)
  2000 Hz | 1.9429 (0.6403) | 1.9143 (0.4365)
  3000 Hz | 3.0286 (0.7944) | 2.7714 (0.5219)
  6000 Hz | 2.2286 (0.4203) | 2.1143 (0.4579)
  8000 Hz | 0.6286 (0.4474) | 1.0000 (0.5266)

3. Secondary Outcome: Tinnitus
Description: Presence of tinnitus was assessed using yes/no question. If tinnitus was reported, perception was assessed using survey.
Time Frame: immediate, repeated measures at 1 hr intervals for 3 hours to measure temporary changes; additional tests at 1 day and 1 week post-exposure.
Population: all participants completing music exposure completed tinnitus surveys.
Measure: Number; unit: participants
Arm/Group | Nutrients | Placebo for Nutrients
Number analyzed (Participants) | 35 | 35
participants | 11 | 6

4. Other Pre Specified Outcome: Distortion Product Otoacoustic Emission (DPOAE) Amplitude - f1+3328 HZ, F2+ 3984 Hz; 30 Minutes
Description: DPOAE amplitude was measured following the audiometric testing completion at approximately 30 minutes post music. Test time was approximate as DPOAE tests began as soon as threshold testing was completed. F1 and F2 frequency pairs included 3328 and 3984 Hz, F1 sound levels started at 65 dB SPL at each frequency, and decreased in 5 dB steps to a level of 25 dB SPL. F2 levels were 10 dB lower than F1 levels. Threshold tests began precisely at 15 min, 1 hr 15 min, 2 hr 15 min, 3 hr 15 min. Threshold tests take approximately 15 min, but the exact duration of testing varies from subject to subject. The OAE testing began as soon as threshold testing completed. Thus, OAE tests began approx. 30 min, 1 hr 30 min, 2 hr 30 min, and 3 hr 30 min post music, but for some it may have been a little bit earlier or a little bit later (i.e., the test may have begun as early as 25 min or as late as 35 min post music, depending on how quickly the subject completed threshold testing).
Time Frame: 15 min
Population: Data for one participant in the placebo group is incomplete.
Measure: Mean (Standard Deviation); unit: decibels (dB)
Groups:
- Nutrients: beta-carotene, vitamins C and E, magnesium
  beta-carotene, vitamins C and E, magnesium: 6 mint-flavored tablets per day, taken once daily
  total daily dose label claim: micronutrient combination of 500 mg vitamin C (magnesium ascorbate), 315 mg magnesium (magnesium citrate, magnesium ascorbate, magnesium stearate), 267 mg vitamin E (d-α-tocopherol acetate), and 18 mg beta carotene.
Arm/Group | Nutrients | Placebo for Nutrients
Number analyzed (Participants) | 35 | 34
decibels (dB)
  f2=3984Hz,f1=65dB,right | 3.9 (9.3) | 6.6 (6.5)
  f2=3984Hz,f1=60dB,right | 0.9 (8.9) | 5.1 (4.6)
  f2=3984Hz,f1=55dB,right | -3.3 (8.8) | 0.5 (6.0)
  f2=3984Hz,f1=50dB,right | -7.8 (9.6) | -4.2 (7.0)
  f2=3984Hz,f1=45dB,right | -13.9 (9.8) | -10.4 (7.7)
  f2=3984Hz,f1=40dB,right | -19.7 (12.8) | -15.6 (8.6)
  f2=3984Hz,f1=35dB,right | -23.8 (8.3) | -21.1 (9.6)
  f2=3984Hz,f1=30dB,right | -25.5 (10.2) | -26.8 (9.7)
  f2=3984Hz,f1=25dB,right | -26.4 (10.6) | -28.0 (11.1)
  f2=3984Hz,f1=65dB,left | 4.4 (8.1) | 4.3 (10.1)
  f2=3984Hz,f1=60dB,left | 1.8 (6.5) | 1.3 (8.5)
  f2=3984Hz,f1=55dB,left | -2.7 (6.8) | -1.3 (7.6)
  f2=3984Hz,f1=50dB,left | -7.0 (7.3) | -7.7 (9.6)
  f2=3984Hz,f1=45dB,left | -13.6 (7.6) | -12.2 (10.2)
  f2=3984Hz,f1=40dB,left | -18.6 (8.7) | -19.2 (10.1)
  f2=3984Hz,f1=35dB,left | -22.1 (12.8) | -23.6 (8.8)
  f2=3984Hz,f1=30dB,left | -30.9 (8.2) | -27.1 (9.0)
  f2=3984Hz,f1=25dB,left | -32.2 (7.7) | -29.8 (8.2)

5. Other Pre Specified Outcome: Threshold Shift at Individual Frequencies, Including 0.25, 0.5, 1, 2, 3, 6, 8, kHz
Time Frame: repeated measures at 1 hr intervals for 3 hours to measure temporary changes; additional tests at 1 day and 1 week post-exposure.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Distortion Product Otoacoustic Emission (DPOAE) Amplitude - Additional Time Measures
Description: DPOAE amplitude was measured following the audiometric testing completion at each of the post-music test times. F1 and F2 frequency pairs included 6656 and 8015 Hz, 5016 and 6000 Hz, 3328 and 3984 Hz, 2484 and 3000 Hz, and 1687 and 2015 Hz. F1 sound levels started at 65 dB SPL at each frequency, and decreased in 5 dB steps to a level of 25 dB SPL. F2 levels were 10 dB lower than F1 levels.
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Distortion Product Otoacoustic Emission (DPOAE) Amplitude - Additional Pairs
Description: Distortion Product Otoacoustic Emission (DPOAE) Amplitude was measured following the audiometric testing completion at approximately 30 minutes post music. F1 and F2 frequency pairs included 6656 and 8015 Hz, 5016 and 6000 Hz, 2484 and 3000 Hz, and 1687 and 2015 Hz. F1 sound levels started at 65 dB SPL at each frequency, and decreased in 5 dB steps to a level of 25 dB SPL. F2 levels were 10dB lower than F1 Levels. Threshold tests began precisely at 15 min, 1 hr 15 min, 2 hr 15 min, 3 hr 15 min. The OAE testing began as soon as threshold testing completed. Threshold tests take approximately 15 min, but the exact duration of testing varies among subjects. Thus, OAE tests began approx. 30 min, 1 hr 30 min, 2 hr 30 min, and 3 hr 30 min post music, but for some it may have been a little bit earlier than for others (i.e., the test may have begun as early as 25 min or as late as 35 min post music, depending on how quickly the subject completed threshold testing).
Time Frame: 15 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: one week
Arm/Group | Nutrients | Placebo for Nutrients
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 2/37 | 5/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nutrients (N=37) | Placebo for Nutrients (N=35)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 2 (2) — includes any report of stomach ache, upset stomach,
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No